CLINICAL TRIAL: NCT04274686
Title: Efficacy of Tegarderm® Placement for Bag Mask Ventilation in the Bearded Patient
Brief Title: Tegarderm® Placement for Bag Mask Ventilation in the Bearded Patient
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention was not seen to be effective on interim analysis
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Neal Gerstein, Professor, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UNMBMVbeard
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Ventilation
Keywords: Tegaderm bandage; Bag mask ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bag-Mask Ventilation with Tegaderm (Experimental): Patients will receive bag-mask ventilation with Tegaderm placement
  Interventions: Device: Tegaderm placement
- Bag-Mask Ventilation without Tegaderm (Active Comparator): Patients will receive bag-mask ventilation without Tegaderm placement
  Interventions: Other: No Tegaderm

INTERVENTIONS:
Device: Tegaderm placement — Placement of perforated Tegaderm bandage over lower face, with diamond-shaped hole aligned with the patient's mouth, for use during bag-mask ventilation
  Arms: Bag-Mask Ventilation with Tegaderm
Other: No Tegaderm — Bag-mask ventilation performed in ordinary fashion, without use of Tegaderm bandage
  Arms: Bag-Mask Ventilation without Tegaderm

SUMMARY:
Difficult Bag Mask Ventilation is well described in the anesthesiology literature, and bearded patients are likely to experience this phenomenon. This study involves application of a large and perforated Tegaderm® across the lower face of the bearded patient to quantify its effectiveness at improving mask ventilation in this anesthetized population.

DETAILED DESCRIPTION:
This study is a prospective crossover trial in bearded patients who will undergo elective or urgent surgery at the main operating rooms of the University of New Mexico Hospital.

It is planned to test the efficacy of the novel bag mask ventilation augmentation technique of placing a large perforated Tegaderm® over the mouth of bearded male patients in order to improve seal after induction of general anesthesia. The perforation is a diamond-shaped hole to be aligned with the patient's mouth. Patients will either start with Tegaderm application or without Tegaderm, and will then cross over to the other condition in order to be their own controls. The primary endpoint is to measure inspiratory and expiratory tidal volumes.

If shown efficacious this intervention would be an easy and cost-effective intervention to improve bag mask ventilation for bearded patients in the operating room and non-operating room environments alike.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with perioral facial hair >5mm in length
* Undergoing elective non-cardiac surgery with planned bag-mask ventilation during anesthesia induction

Exclusion Criteria:

* Known allergy to Tegaderm product and/or its adhesive
* Emergency surgery
* Active or unstable cardiac disease
* ASA (American Society of Anesthesiologists) physical status ≥4
* External or internal active airway obstruction from tumor, abscess, or laryngeal edema
* Organic or non-organic oropharyngeal anatomical defects including history of radiation treatment to the neck
* Moderate to severe acute and chronic restrictive or obstructive lung diseases, e.g. chronic obstructive pulmonary disease, asthma, etc.
* Requirement for rapid sequence intubation, or known aspiration risk
* Cervical spine injury
* Previously documented difficult mask ventilation or intubation
* BMI ≥50
* Vulnerable populations: children, prisoners, pregnant patients, cognitively impaired adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Gerstein, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerstein NS, Braude DA, Petersen TR, Goumas A, Fish AC, Panikkath PV. Use of Transparent Film Dressing to Facilitate Mask Ventilation in Bearded Patients. J Emerg Med. 2024 Feb;66(2):163-169. doi: 10.1016/j.jemermed.2023.07.008. Epub 2023 Jul 20. PMID 38238230

RESULTS

PARTICIPANT FLOW:
Groups:
- Tegaderm-First Group: Patients will first receive bag-mask ventilation with a perforated Tegaderm sheet in place, and then with the sheet removed
- Without-Tegaderm First Group: Patients will first receive bag-mask ventilation as in usual practice without a Tegaderm sheet in place, and then will receive bag-mask ventilation with a perforated Tegaderm sheet covering the lower face and beard
Period: Overall Study
Arm/Group | Tegaderm-First Group | Without-Tegaderm First Group
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants in the study
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25
Beard Length [Count of Participants; unit: Participants]
  5 mm | 8
  5-9 mm | 3
  1 cm | 6
  >1 cm | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Air Leakage During Bag-mask Ventilation
Description: Leakage defined as difference in inspired and expired tidal volumes during bag-mask ventilation, as a percentage of inspired tidal volume.
Time Frame: <5 minutes
Measure: Mean (Standard Deviation); unit: percentage of inspired tidal volume
Groups:
- Bag-mask Ventilation With Tegaderm Placement: Bag-mask ventilation in study condition with perforated Tegaderm sheet placed over lower face and beard
- Bag-mask Ventilation Without Tegaderm Placement: Bag-mask ventilation in control condition with mask placed directly over face and beard, as in usual practice, with no Tegaderm sheet
Arm/Group | Bag-mask Ventilation With Tegaderm Placement | Bag-mask Ventilation Without Tegaderm Placement
Number analyzed (Participants) | 24 | 24
percentage of inspired tidal volume | 47.6 (26.2) | 45.7 (20.4)
Statistical Analysis 1: Comparison: Bag-mask Ventilation With Tegaderm Placement vs Bag-mask Ventilation Without Tegaderm Placement; Null hypothesis: No difference in percent air leakage; Test type: Superiority; p = 0.667, Paired t-test; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-7.0 to 10.7]

2. Secondary Outcome: Resistance
Description: Airflow resistance during bag-mask ventilation
Time Frame: <5 minutes
Measure: Mean (Standard Deviation); unit: cm H2O/L/s
Arm/Group | Bag-mask Ventilation With Tegaderm Placement | Bag-mask Ventilation Without Tegaderm Placement
Number analyzed (Participants) | 24 | 24
cm H2O/L/s | 8.83 (5.57) | 7.73 (3.69)
Statistical Analysis 1: Comparison: Bag-mask Ventilation With Tegaderm Placement vs Bag-mask Ventilation Without Tegaderm Placement; Test type: Superiority; p = 0.218, Paired t-test; Mean Difference (Final Values) = 1.10, 95% CI 2-sided [-0.70 to 2.90]

3. Secondary Outcome: Peak Inspiratory Pressure
Description: Maximum air pressure observed during bag-mask ventilation
Time Frame: <5 minutes
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Bag-mask Ventilation With Tegaderm Placement | Bag-mask Ventilation Without Tegaderm Placement
Number analyzed (Participants) | 24 | 24
cm H2O | 19.3 (1.6) | 19.4 (1.3)
Statistical Analysis 1: Comparison: Bag-mask Ventilation With Tegaderm Placement vs Bag-mask Ventilation Without Tegaderm Placement; Test type: Superiority; p = 0.455, Paired t-test; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.5 to 0.2]

ADVERSE EVENTS:
Time Frame: 10 minutes
Groups:
- Bag-mask Ventilation With Tegaderm Placement: Bag-mask ventilation performed with perforated Tegaderm sheet placed over the lower face and beard
- Bag-mask Ventilation Without Tegaderm Placement: Bag-mask ventilation performed as in usual practice, with mask placed directly over lower face and beard
Arm/Group | Bag-mask Ventilation With Tegaderm Placement | Bag-mask Ventilation Without Tegaderm Placement
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT04274686/Prot_SAP_002.pdf
  • Informed Consent Form (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT04274686/ICF_003.pdf